CLINICAL TRIAL: NCT06630429
Title: A Pilot Study of Blood-Based Biomarkers for Response to Immune Checkpoint Inhibitors
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Dwight Owen, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-20001
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer; Renal Cell Carcinoma (RCC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Includes patients with Stage IB-IV NSCLC receiving treatment with immune checkpoint inhibitors either alone or in combination with chemotherapy.
  Interventions: Other: Biospecimen Collection
- Cohort B: Includes patients with metastatic RCC receiving first line combination with nivolumab and ipilimumab.
  Interventions: Other: Biospecimen Collection

INTERVENTIONS:
Other: Biospecimen Collection — Undergo collection of blood and stool samples

SUMMARY:
A pilot study evaluating baseline and on-treatment changes in tumor fraction (TFx) in peripheral blood in patients with NSCLC and RCC being treated with checkpoint inhibitor therapy as part of standard of care. The primary objective of the study is to determine whether baseline TFx can be reliably predicted in patients with NSCLC and RCC and if changes can be detected during treatment that may correlate with response. Exploratory analyses will be completed to assess the potential roles of cachexia-associated inflammation, tumor-associated increases in glucocorticoid secretion, and ketosis/ketogenesis in both elevated mAb clearance and in response to ICI therapy. Measurements will include circulating IL-6 and other cytokine levels, glucocorticoid levels, ketone levels and stool analysis for assessment of gut microbiome.

DETAILED DESCRIPTION:
Primary objective:

The primary objective of this protocol is to establish whether TFx can be reliably measured in patients with NSCLC and RCC undergoing treatment with ICI

Secondary objectives:

* To incorporate and evaluate relationships among other known risk factors for cachexia relative to ICI therapy pharmacokinetics and clinical outcomes (to include baseline and longitudinal measures of body weight, body composition determinations via L3 CT scans, and albumin for cachexia, and baseline ICI mAb clearance and changes in clearance over time for PK).
* To determine whether detected changes in TFx can be appreciated during treatment and whether these changes are associated with clinical benefit by RECIST v1.1, progression free survival (PFS) and overall survival (OS).

Exploratory Objectives:

* To determine potential roles of cachexia-associated inflammation, tumor-associated increases in glucocorticoid secretion, and ketosis/ketogenesis in both elevated mAb clearance and in response to ICI therapy (by RECIST 1.1, PFS, and OS)

  * This includes measurement of cytokines and other signaling markers, including, but not limited to IL-6, Interferon-γ and TGF-β
  * Endogenous glucocorticoids and ketones
  * Soluble PD-L1
  * Ki-67+PD-1+CD8+ T cells, Treg cells, and PBMC analysis for measurement of expression of FcRn
* To quantify the performance of a modifiable biomarker - the gut microbiome - to use as a predictive indicator of clinical benefit in lung cancer patients who receive randomized treatment combinations.
* To determine whether TFx changes differ by stage of cancer or setting of ICI therapy in NSCLC 11
* To compare peripheral blood changes in inflammation including CD8+ T Cells and Treg

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥ 18 years
2. Cohort A will include patients with confirmed diagnosis of all non-small cell lung cancer (NSCLC) histologies including adenocarcinoma, squamous cell, adenosquamous, sarcomatoid/pleomorphic, and poorly differentiated/NOS, as well as patients diagnosed with malignant pleural mesothelioma. Cohort B will include patients with confirmed diagnosis of RCC (clear cell or any non-clear cell histology) receiving first treatment with immunotherapy alone or in combination therapy for metastatic disease or as adjuvant or neoadjuvant therapy.
3. Patients planned for standard of care treatment with immune checkpoint inhibitors (ICIs, see appendix 3 for list) either as monotherapy or in combination therapy.
4. Scheduled for imaging every 6 to 12 weeks for stage IV NSCLC and RCC as is standard of care per NCCN guidelines.
5. Able to read, understand, and provide written informed consent.

g. Willing to provide blood specimen and stool samples for research studies as outlined in the calendar h. ECOG performance status 0-2 i. Life expectancy ≥ 3 months

Exclusion Criteria:

1. Individuals <18 years of age
2. Patients who have received previous immune checkpoint inhibitor therapy.
3. Unable or unwilling to provide consent.
4. Other malignancy requiring active ongoing treatment with systemic therapy (excluding hormonal therapy).
5. Women who are known to be pregnant are excluded. However no additional pregnancy testing out of what would be recommended prior to initiating anti-cancer therapy will be performed solely for this study.
6. Patients currently participating in an interventional or therapeutic clinical trial involving the use of active anti-cancer therapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects receiving care at The Ohio State University Comprehensive Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with tumor fraction change | From enrollment up to 12 months
  The primary outcome is the percentage of patients having >5% change (better or worse) in tumor fraction during the first two cycles. With 90 patients having detectable tumor fraction, the % of patients having >5% change in tumor fraction can be estimated with a 95% confidence interval of ±10%. Assuming the response rate of 30%, 27 responders will provide at least 80% power to detect an effect size of 0.5 standard deviations reduction of tumor fraction from baseline to treatment by cycle 3 at significance level of 0.05, based on a one-sided paired t-test. If the response rate is higher, a smaller reduction can be detected.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: Related Info — http://cancer.osu.edu